CLINICAL TRIAL: NCT03529799
Title: Examining Disparity Driven Vergence as a Potential Diagnostic Test for Mild Traumatic Brain Injury (mTBI)
Brief Title: Disparity Driven Vergence in Mild Traumatic Brain Injury (mTBI)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: University of Miami (Other)
Collaborators: Neurolign (Industry)
Responsible Party: Principal Investigator, Michael E. Hoffer, Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20180058
Record Dates: First submitted 2018-04-24; First posted 2018-05-18 (Actual); Results first posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Mild Traumatic Brain Injury
Keywords: mTBI; TBI; brain injury; concussion
MeSH Terms: conditions — Brain Concussion; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Injured Participants (Experimental): Participants with mild traumatic brain injury (mTBI) tested using the I-PAS goggles
  Interventions: Device: I-PAS Goggles
- Uninjured Participants (Active Comparator): Participants with no mild traumatic brain injury (mTBI) tested using the I-PAS goggles
  Interventions: Device: I-PAS Goggles

INTERVENTIONS:
Device: I-PAS Goggles — Portable, head-mounted display goggle system with integrated eye capture technology

SUMMARY:
This study aims to determine the validity and safety of disparity driven vergence using a portable goggle system (I-PAS) using a pseudorandom ternary sequence of frequencies for testing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* Both females and males

Exclusion Criteria:

* Central processing disorder
* Impaired vision without corrective lenses (max 20/60 uncorrected)
* Moderate to severe hearing loss (>55 decibels (dB) pure tone audiometry (PTA), <50% word identification)
* Vestibular disorder except for patients recruited for subjects recruited with a history of mild traumatic brain injury to compare to normal participants
* History of ear surgery other than myringotomy with or without tube placement
* Pregnant women
* Prisoners
* Adults unable to consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hoffer, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Injured Participants | Uninjured Participants
Started | 14 | 26
Completed | 14 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Injured Participants | Uninjured Participants | Total
Number analyzed (Participants) | 14 | 26 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (16.9) | 33.4 (9.7) | 34.05 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 19 | 27
  Male | 6 | 7 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucsian: Hispanic | 8 | 16 | 24
  Caucsian: Caucasian | 4 | 6 | 10
  Caucsian: Other | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Pseudorandom Ternary Sequence of Frequency
Description: Pseudorandom Ternary Sequence of Frequency (reported in Hertz) will be measured via mergence testing using the IPAS goggles.
Time Frame: 15 minutes
Population: All participants
Measure: Median (Standard Deviation); unit: Hertz
Arm/Group | Injured Participants | Uninjured Participants
Number analyzed (Participants) | 14 | 26
Hertz | 0.07 (0.69) | 0.1 (0.54)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Injured Participants | Uninjured Participants
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/26
Other Adverse Events (participants affected / at risk) | 0/14 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/99/NCT03529799/Prot_SAP_000.pdf